CLINICAL TRIAL: NCT05828563
Title: Immunological Indices and Infections Among Pesticide Applicators in Sohag Governorate
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Yara Mohamed Ahmed, DEMONSTRATOR, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh-Med-23-4-05MS
Record Dates: First submitted 2023-04-13; First posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Pesticide Adverse Reaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pesticide applicators (Active Comparator): This group contain cases
  Interventions: Diagnostic Test: Blood sample test
- control (Active Comparator): control group
  Interventions: Diagnostic Test: Blood sample test

INTERVENTIONS:
Diagnostic Test: Blood sample test — Blood sample will be taken to determine immunological indices

SUMMARY:
The human body gets exposure to pesticides either directly or indirectly. By using pesticides on crops, humans come in direct contact with them and they affect the heaith

Immune system is the first defense line against pathogenic organisms; however, it is altered by the vulnerable environmental factors such as pesticides, which can cause structural or functional alterations in humoral or cell mechanisms (nonspecific or adaptive) of the immune response which lead to an increase in the susceptibility to infections

ELIGIBILITY:
Inclusion Criteria:

1. pesticide applicators
2. Age ;20-60 years
3. Exposure to pesticides for more than 3 months

Exclusion Criteria:

* Subjects have recent severe trauma or surgery or recent infections

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
immunlogical indices | 12 months
  immunoglobulins (IgG ,IgE)

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hadnagy W, Leng G, Sugiri D, Ranft U, Idel H. Pyrethroids used indoors--immune status of humans exposed to pyrethroids following a pest control operation--a one year follow-up study. Int J Hyg Environ Health. 2003 Mar;206(2):93-102. doi: 10.1078/1438-4639-00201. PMID 12708230
- [Background] Kalyabina VP, Esimbekova EN, Kopylova KV, Kratasyuk VA. Pesticides: formulants, distribution pathways and effects on human health - a review. Toxicol Rep. 2021 Jun 6;8:1179-1192. doi: 10.1016/j.toxrep.2021.06.004. eCollection 2021. PMID 34150527
- [Background] Zhang W, Lin Z, Pang S, Bhatt P, Chen S. Insights Into the Biodegradation of Lindane (gamma-Hexachlorocyclohexane) Using a Microbial System. Front Microbiol. 2020 Mar 27;11:522. doi: 10.3389/fmicb.2020.00522. eCollection 2020. PMID 32292398